CLINICAL TRIAL: NCT03007160
Title: A Randomized, Blank Controlled, Multicenter Clinical Trial of the Effection of Potassium Citrate Extended-release Tablets on Urolithiasis Formation or Recurrence
Brief Title: A Study on the Effection of Potassium Citrate Extended-release Tablets on Urolithiasis Formation or Recurrence
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dawnrays Pharmaceutical (Holdings) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAWNRAYS101
Record Dates: First submitted 2016-12-13; First posted 2017-01-02 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Potassium Citrate Extended-release Tablets
  Interventions: Drug: Potassium Citrate Extended-release Tablets
- Blank control group (No Intervention): Subjects do not take the investigational product

INTERVENTIONS:
Drug: Potassium Citrate Extended-release Tablets — Daily 3.24g, Po ,Tid, each 1.08g/tablets
  Other Names: Juyuansuanjia Huanshi Pian
  Arms: Experimental group

SUMMARY:
Assess the efficacy and safety of potassium citrate extended-release tablets on Urolithiasis formation or recurrence.

DETAILED DESCRIPTION:
This study takes "Rate of stone recurrence" as primary outcome measure, by random, blank control, and multicenter clinical trial design method, assess the efficacy and safety of potassium citrate extended-release tablets on Urolithiasis formation or recurrence, provide evidence for drug re-registration, and observe its efficacy on Urinary calculi such as renal tubular acidosis with calcium stone, and uric acid stones with or without calcium stone, urinary tract stone of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper urinary tract calculi surgery and/or ESWL within 3 months；
* Stone free or had residual stone fragments with a less than 4 mm diamete；
* 18-70 years of age; the gender is not limited；
* Agree to take effective contraceptive measures during the study period, and female of childbearing age whose pregnancy test is negative；
* Subjects with no mental illness and language dysfunction, can understand the situation of the study and have signed informed consent.

Exclusion Criteria:

* Patients with infectious stones, medical stones and urinary tract obstruction；
* Patients with hyperkalemia (K+>5.5mmol/L) (or patients with factors or disease that can cause hyperkalemia), because the further increase in blood potassium can lead to cardiac arrest. These factors include disease or strenuous exercise, chronic renal failure, uncontrolled diabetes, acute dehydration, excessive, adrenal insufficiency, extensive tissue failure. Patients who takes potassium sparing diuretics (such as triamterene, spironolactone, amiloride)；
* Patients with gastrointestinal disorders, such as peptic ulcer, severe vomiting, diarrhea, delayed gastric emptying, intestinal obstruction, etc.；
* Combined with cardiovascular, liver, kidney, hematopoietic system, such as severe primary disease, or known to affect the survival of serious diseases (such as cancer or AIDS), or patients with with disabilities mentally or legally；
* Patients with renal insufficiency (1.2 times the upper limit of the normal value of serum creatinine and urea nitrogen)；
* The recent (within 6 months) with family planners；
* Allergic to this product；
* To participate in other clinical trials in the past three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2001 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Urolithiasis recurrence | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Time of stone recurrence | through study completion, an average of 1 year
The changes of urine citric acid content compared with baseline | through study completion, an average of 1 year
The changes of Urine pH value compared with baseline | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhangqun YE, M.D., Principal Investigator — Tongji Hospital
Locations (6):
- China (6):
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan No.1 Hospital（Wuhan Integrated TCM & Western Medicine Hospital）, Wuhan, Hubei
  - Shanghai Ninth People's Hospital,Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sfoungaristos S, Gofrit ON, Yutkin V, Pode D, Duvdevani M. Prevention of renal stone disease recurrence. A systematic review of contemporary pharmaceutical options. Expert Opin Pharmacother. 2015 Jun;16(8):1209-18. doi: 10.1517/14656566.2015.1037740. Epub 2015 Apr 16. PMID 25881654
- [Background] Soygur T, Akbay A, Kupeli S. Effect of potassium citrate therapy on stone recurrence and residual fragments after shockwave lithotripsy in lower caliceal calcium oxalate urolithiasis: a randomized controlled trial. J Endourol. 2002 Apr;16(3):149-52. doi: 10.1089/089277902753716098. PMID 12028622
- [Background] Lee YH, Huang WC, Tsai JY, Huang JK. The efficacy of potassium citrate based medical prophylaxis for preventing upper urinary tract calculi: a midterm followup study. J Urol. 1999 May;161(5):1453-7. PMID 10210371
- [Background] Fabris A, Lupo A, Bernich P, Abaterusso C, Marchionna N, Nouvenne A, Gambaro G. Long-term treatment with potassium citrate and renal stones in medullary sponge kidney. Clin J Am Soc Nephrol. 2010 Sep;5(9):1663-8. doi: 10.2215/CJN.00220110. Epub 2010 Jun 24. PMID 20576821
- [Background] Bartoletti R, Cai T, Mondaini N, Melone F, Travaglini F, Carini M, Rizzo M. Epidemiology and risk factors in urolithiasis. Urol Int. 2007;79 Suppl 1:3-7. doi: 10.1159/000104434. PMID 17726345